CLINICAL TRIAL: NCT02144909
Title: Partners in Care With Semi-Structured Support Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Claire Townsend, Clinical Research Specialist, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHS-21514; U54MD007584 (NIH)
Record Dates: First submitted 2013-11-15; First posted 2014-05-22 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes self management; support group; semi structured support group
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partners in Care with Semi-Structured Support Group (Experimental): Partners in Care with Semi-Structured Support Group: participants will receive the Partners in Care intervention followed by 6 semi-structured support groups, conducted every other week for 3 months. Half of the support groups will be conducted by professionals with diabetes specific knowledge, e.g., pharmacists, physicians, nutritionists. While the other half will be conducted by the trained diabetes self-management facilitator.
  Interventions: Behavioral: Partners in Care with Semi-Structured Support Group
- Partners in Care Standard Follow-up (No Intervention): Participants will receive the Partners in Care intervention followed by monthly healthy lifestyle tips related to diabetes self-management

INTERVENTIONS:
Behavioral: Partners in Care with Semi-Structured Support Group
  Arms: Partners in Care with Semi-Structured Support Group

SUMMARY:
The investigators are conducting a feasibility study using a randomized controlled trial (RCT) design in which participants will receive the Partners in Care (PIC) diabetes self-management intervention and then be randomized to either semi-structured social support or a standard follow-up control group. Participants in the support groups will receive a culturally-tailored, semi-structured social support program delivered in a community setting by trained community peer educators and other health professionals (e.g., pharmacist). The investigators believe that the addition of a semi-structured social support component as a supplement to an evidence-based diabetes self-management intervention will improve diabetes self-care maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Native Hawaiian, Filipino, or other Pacific Islander ethnic background
* Adults age >18 years of age
* English-speaking
* Physician-diagnosed type 2 diabetes
* Baseline hemoglobin A1c >8%

Exclusion Criteria:

* Survival less than 6 months
* Planning to move out of the community during the intervention study period
* Pregnancy
* Any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (i.e., major psychiatric illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline hemoglobin a1c at 3 months and at 6 months | baseline, 3 months, 6 months
Change from Baseline diabetes management functioning as measured by the Problem Areas in Diabetes questionnaire at 3 months and 6 months | baseline, 3 months, 6 months
  The PAID is a 20-item instrument that assesses the physical and social functioning of patients as well as their perceived level of mental and emotional well-being specific to living with diabetes.

SECONDARY OUTCOMES:
Change from Baseline blood pressure at 3 months and 6 months | baseline, 3 months, 6 months
Change from Baseline Total Cholesterol (including HDL and LDL) and triglycerides at 3 months and 6 months | baseline, 3 months, 6 months
  Total Cholesterol (including HDL and LDL) and triglycerides will be measured with the Cholestech LDX analyzer
Change from Baseline weight in kg at 3 months and 6 months | baseline, 3 months, 6 months

OTHER OUTCOMES:
Change from Baseline reported diabetes self-care activities as measured by the Summary of Diabetes Self-Care Activities questionnaire at 3 months and 6 months | baseline, 3 months, 6 months
Change from Baseline reported amount of support as measured a questionnaire at 3 months and 6 months | baseline, 3 months, 6 months
Change from Baseline amount of physical activity as measured a questionnaire at 3 months and 6 months | baseline, 3 months, 6 months
Change from Baseline dietary patterns as a questionnaire at 3 months and 6 months | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kula no na Po'e Hawai'i, Honolulu, Hawaii
  - Ke Ola Mamao, Honolulu, Hawaii
  - Kokua Kalihi Valley, Honolulu, Hawaii

REFERENCES:
- [Background] Sinclair KA, Makahi EK, Shea-Solatorio C, Yoshimura SR, Townsend CK, Kaholokula JK. Outcomes from a diabetes self-management intervention for Native Hawaiians and Pacific People: Partners in Care. Ann Behav Med. 2013 Feb;45(1):24-32. doi: 10.1007/s12160-012-9422-1. PMID 23086589
- [Derived] Townsend CK, Dillard A, Hosoda KK, Maskarinec GG, Maunakea AK, Yoshimura SR, Hughes C, Palakiko DM, Kehauoha BP, Kaholokula JK. Community-Based Participatory Research Integrates Behavioral and Biological Research to Achieve Health Equity for Native Hawaiians. Int J Environ Res Public Health. 2015 Dec 22;13(1):ijerph13010004. doi: 10.3390/ijerph13010004. PMID 26703660